CLINICAL TRIAL: NCT00646841
Title: The Effects of Doxazosin Gastrointestinal Therapeutic System (GITS) on Ambulatory Blood Pressure and Cardiovascular Risk Factors in Uncontrolled Hypertensives on Drug Therapy
Brief Title: Effects of Doxazosin Gastrointestinal Therapeutic System on Ambulatory Blood Pressure and Cardiovascular Risk Factors in Uncontrolled Hypertensive Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A0351051
Record Dates: First submitted 2008-03-26; First posted 2008-03-31 (Estimated); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Hypertension
Keywords: Essential hypertension, doxazosin, ambulatory blood pressure monitoring
MeSH Terms: conditions — Hypertension; Essential Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental)
  Interventions: Drug: Doxazosin gastrointestinal therapeutic system (GITS)

INTERVENTIONS:
Drug: Doxazosin gastrointestinal therapeutic system (GITS) — 4 mg/day, and was titrated, if necessary, to 8 mg/day at Week 3 (Visit 5) or Week 5 (Visit 6).

SUMMARY:
The primary objective was to determine the effects of the Gastrointestinal Therapeutic System (GITS) formulation of Doxazosin when used in combination therapy with the 5 major classes of antihypertensive agents as measure by 24-hour diastolic blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* Eligible subjects were males or females ≥18 years of age with a diagnosis of primary essential hypertension and currently taking 1 or 2 individual antihypertensive agents
* Dosing for entry antihypertensive medication was at the accepted efficacious dose or the maximum tolerated dose and had to be stable for at least 4 weeks prior to study entry
* Subjects were required to have clinic sitting DBP ≥95 and ≤110 mmHg and SBP ≥140 and ≤180 mmHg as an average of 3 readings on their current antihypertensive therapy at visits 1 and 2

Exclusion Criteria:

Exclusion criteria included, but were not limited to:

* Subjects taking antihypertensive medications for other indications (i.e. arrhythrma, unstable angina, CHF, etc.)
* Orthostatic hypotension, defined as a decrease of at least 20 mmHg systolic or 1OmmHg diastolic pressure between sitting and standing blood pressures after 2 rmnutes, or known fluid depletion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2003-02; Primary Completion 2004-02 (Actual); Study Completion 2004-02 (Actual)

PRIMARY OUTCOMES:
To determine the effects of Doxazosin Gastrointestinal Therapeutic System (GITS) 4 or 8mg/day on mean 24-hour diastolic ambulatory blood pressure (ABP) when used in combination therapy in subjects with uncontrolled essential hypertension. | 11 weeks

SECONDARY OUTCOMES:
Serum lipid levels (total cholesterol [TC], HDL cholesterol, calculated LDL cholesterol, triglycerides, calculated HDL/TC ratio) | 9 weeks
HgbA1C | 9 weeks
24-hour systolic ABP and 24-hour ambulatory heart rate | 9 weeks
daytime and nighttime (2200 to 0600 hours) ABP and ambulatory heart rate | 9 weeks
Sitting and standing clinic blood pressure (BP) and heart rate | 9 weeks
24-hour ABP smoothness index | 9 weeks
24-hour ABP and ambulatory heart rate between 24 hours (Week 9) and 48 hours (Week 9+1 day) after final dose of Doxazosin GITS | 9 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (7):
- Italy (3):
  - Pfizer Investigational Site, Brescia
  - Pfizer Investigational Site, Monza (Milan)
  - Pfizer Investigational Site, Padua
- Spain (2):
  - Pfizer Investigational Site, Palamós, Gerona
  - Pfizer Investigational Site, Madrid
- Pfizer Investigational Site, London, United Kingdom
- Pfizer Investigational Site

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0351051&StudyName=Effects%20of%20Doxazosin%20Gastrointestinal%20Therapeutic%20System%20on%20Ambulatory%20Blood%20Pressure%20and%20Cardiovascular%20Risk%20Factors%20in%20Uncontrolled%20Hyperten